CLINICAL TRIAL: NCT01154868
Title: Clinical and Histological Evaluation of Healos® for Alveolar Ridge Augmentation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor withdrew funding of study.
Sponsor: William Giannobile (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor-Investigator, William Giannobile, William Giannobile, D.D.S., D.Med.Sc., University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00035937
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Dental Implantation
MeSH Terms: interventions — Alveolar Ridge Augmentation; Healos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healos (Other)
  Interventions: Procedure: Alveolar ridge augmentation

INTERVENTIONS:
Procedure: Alveolar ridge augmentation — Under local anesthesia, full-thickness mucoperiosteal flaps will be elevated, followed by degranulation, and collection of all clinical measurements. Crestal and vertical releasing cuts will be performed using diamond-coated discs on the edentulous ridge in need of augmentation. A sequence of bone chisels and osteotomes will be used to split the alveolar ridge in half until a desirable width for implant placement is achieved. Healos® will then be inserted between both osseous plates. Fixation screws will be used as needed to stabilize the expanded alveolar ridge. Collagen barrier membranes (Ossix Plus) will be used to cover the osseous wound. Flaps will be approximated to achieve primary wound closure.
  Other Names: Healos

SUMMARY:
The purpose of this study is to document and evaluate how a bone graft material (Healos®) can help rebuild bone width. Dental implants can only be placed when enough bone is found and this bone graft may help to rebuild bone width for dental implant placement. The ultimate goal of this study is to evaluate how this graft material can help bone healing.

ELIGIBILITY:
Inclusion Criteria:

* age 21 and older
* 2-4 ADJACENT maxillary front teeth missing
* require ridge augmentation and dental implant
* nonsmoker for at least 6 months
* willing to follow oral hygiene instruction and other study instruction
* able to read, understand and sign informed consent

Exclusion Criteria:

* Residual upper jaw bone equal to or narrower than 3mm.
* Insufficient gum tissue to obtain wound closure after surgery.
* Clinically significant or unstable (as defined by the investigators) systemic diseases affecting bone or soft tissue growth; or other kidney, liver, heart, thyroid, blood, autoimmune or acute infectious diseases that makes interpretation of the data more difficult
* A history of head & neck radiation treatment due to certain medical conditions.
* Taking steroids, tetracycline or tetracycline analogs, bone therapeutic levels of fluorides, bisphosphonates, medications affecting bone turnover, antibiotics for >7 days or any investigational drug
* Pregnancy or become pregnant during the length of the study
* Wearing removable partial dentures that may put pressure over the area where the bone graft will be placed.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
horizontal (width) bone gain or loss in millimeters. | 18 weeks

SECONDARY OUTCOMES:
radiographic bone changes measured using computer tomography | 18 weeks
percentage of new bone formation in the alveolar bone core biopsies. | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Giannobile, DDS, DMedSc, Principal Investigator — University of Michigan
Locations (1):
- Michigan Center for Oral Health Research, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Engler WO, Ramfjord SP, Hiniker JJ. Healing following simple gingivectomy. A tritiated thymidine radioautographic study. I. Epithelialization. J Periodontol. 1966 Jul-Aug;37(4):298-308. doi: 10.1902/jop.1966.37.4.298. No abstract available. PMID 4287364
- [Background] Ramfjord SP, Engler WO, Hiniker JJ. A radioautographic study of healing following simple gingivectomy. II. The connective tissue. J Periodontol. 1966 May-Jun;37(3):179-89. doi: 10.1902/jop.1966.37.3.179. No abstract available. PMID 4956575
- [Background] HURLEY LA, STINCHFIELD FE, BASSETT AL, LYON WH. The role of soft tissues in osteogenesis. An experimental study of canine spine fusions. J Bone Joint Surg Am. 1959 Oct;41-A:1243-54. No abstract available. PMID 13852565
- [Background] MURRAY G, HOLDEN R, ROSCHLAU W. Experimental and clinical study of new growth of bone in a cavity. Am J Surg. 1957 Mar;93(3):385-7. doi: 10.1016/0002-9610(57)90827-9. No abstract available. PMID 13403056
- [Background] Buser DA, Tonetti M. Clinical trials on implants in regenerated bone. Ann Periodontol. 1997 Mar;2(1):329-42. doi: 10.1902/annals.1997.2.1.329. PMID 9151565
- [Background] Scipioni A, Calesini G, Micarelli C, Coppe S, Scipioni L. Morphogenic bone splitting: description of an original technique and its application in esthetically significant areas. Int J Prosthodont. 2008 Sep-Oct;21(5):389-97. PMID 18950058
- [Background] Simion M, Baldoni M, Zaffe D. Jawbone enlargement using immediate implant placement associated with a split-crest technique and guided tissue regeneration. Int J Periodontics Restorative Dent. 1992;12(6):462-73. PMID 1298734
- [Background] Engelke WG, Diederichs CG, Jacobs HG, Deckwer I. Alveolar reconstruction with splitting osteotomy and microfixation of implants. Int J Oral Maxillofac Implants. 1997 May-Jun;12(3):310-8. PMID 9197095
- [Background] Coatoam GW, Mariotti A. The segmental ridge-split procedure. J Periodontol. 2003 May;74(5):757-70. doi: 10.1902/jop.2003.74.5.757. PMID 12816307
- [Background] Basa S, Varol A, Turker N. Alternative bone expansion technique for immediate placement of implants in the edentulous posterior mandibular ridge: a clinical report. Int J Oral Maxillofac Implants. 2004 Jul-Aug;19(4):554-8. PMID 15346753
- [Background] Neen D, Noyes D, Shaw M, Gwilym S, Fairlie N, Birch N. Healos and bone marrow aspirate used for lumbar spine fusion: a case controlled study comparing healos with autograft. Spine (Phila Pa 1976). 2006 Aug 15;31(18):E636-40. doi: 10.1097/01.brs.0000232028.97590.12. PMID 16915079